CLINICAL TRIAL: NCT04424771
Title: PTSD in Health Workers During COVID-19 Pandemia
Brief Title: Post-traumatic Stress Disease in Health Workers During COVID-19 Pandemia
Status: Completed | Type: Observational
Sponsor: Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia (Other)
Responsible Party: Principal Investigator, Simone Ferrero, Principal investigator, Piazza della Vittoria 14 Studio Medico - Ginecologia e Ostetricia
Other Study IDs: PTSD-COVID-19
Record Dates: First submitted 2020-06-07; First posted 2020-06-11 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: COVID; Post Traumatic Stress Disorder
Keywords: COVID-19
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; COVID-19 | interventions — Maslach Burnout Inventory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health workers: They include doctors, nurses, techinicians, biologists and other non technical inhospital workers
  Interventions: Behavioral: Maslach Burnout Inventory (MBI)

INTERVENTIONS:
Behavioral: Maslach Burnout Inventory (MBI) — The Maslach Burnout Inventory is an introspective psychological inventory consisting of 22 items pertaining to occupational burnout.

SUMMARY:
The purpose of the questionnaire is to find risk factors for the development of post-traumatic stress disease (PTSD) in health workers during COVID-19 pandemy.

ELIGIBILITY:
Inclusion Criteria:

* workers in health services, including phisicians, nurses, inhospital technicians and biologists

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consisted of workers in health services.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with diagnosis of PTSD. | Through study completion, an average of 1 months
  PTSD consists in job burnout, including emotional exhaustion, depersonalization, and personal accomplishment.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Ospedale Perrino Asl Brindisi, Brindisi
  - Piazza della Vittoria 14 Studio medico - Ginecologia e Ostetricia, Genoa

IPD SHARING:
Plan to Share IPD: Undecided